CLINICAL TRIAL: NCT03445013
Title: A Phase 1b Multi-Center, Double-Blind, Randomized, Vehicle-Controlled Study Assessing the PK, Pharmacodynamics, Safety, and Tolerability of SB414 in Subjects With Psoriasis
Brief Title: A Study Assessing the PK, PD, Safety, and Tolerability of SB414 in Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novan, Inc. (Industry)
Collaborators: Novella Clinical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NI-PS101
Record Dates: First submitted 2018-01-31; First posted 2018-02-26 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — berdazimer sodium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SB414 6% (Experimental): SB414 6% topically twice daily
  Interventions: Drug: SB414 6%
- Vehicle Cream (Placebo Comparator): Vehicle Cream topically twice daily
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: SB414 6% — Twice daily
  Other Names: NVN1000
  Arms: SB414 6%
Drug: Vehicle — Vehicle Comparator
  Other Names: Placebo
  Arms: Vehicle Cream

SUMMARY:
The objectives of this study are to assess the pharmacokinetics, pharmacodynamics, safety, and tolerability of SB414 in subjects with mild to moderate plaque psoriasis.

DETAILED DESCRIPTION:
This is a phase 1b, multi-center, double-blind, randomized, vehicle-controlled study to be conducted in approximately 36 adult subjects with mild to moderate chronic plaque psoriasis. After obtaining informed consent, subjects will be randomized to active or vehicle treatment arms. Subjects will apply the study product (SB414 6% or Vehicle cream) twice daily to all affected areas of psoriasis on the trunk and/or extremities for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female, 18-70 years old, and in good general health;
* Have a clinical diagnosis of stable chronic plaque psoriasis of mild to moderate severity based on the PSGA, involving 2-15% BSA (excluding the scalp/face), present for > 6 months;
* Must have at least 2 target plaques on trunk and/or extremities at least 5 cm2 with a TPSS > 5 and thickness sub-score > 2. Target plaques cannot be located on the groin, hands, feet, neck, face, elbows, knees, ankles or scalp;
* Be willing to not use any other systemic agents used to treat psoriasis or apply any other topical products (medicated or over-the-counter) to the treatment sites on the trunk and/or extremities during the study;
* Women of childbearing potential (WOCBP) must have a negative UPT prior to randomization and must agree to use an effective method of birth control during the study and for 30 days after their final study visit.

Exclusion Criteria:

* Have inverse (i.e.: axillae, groin) or facial psoriasis only, erythrodermic psoriasis, guttate psoriasis, pustular psoriasis, drug-induced psoriasis, and /or psoriatic arthritis requiring treatment with disease modifying antirheumatic drugs (DMARDs);
* Concurrent or recent use of topical or systemic medications without a sufficient washout period;
* Are immunocompromised, including those who are known HIV positive or received immunosuppressive treatment within the past 6 months;
* Female subjects who are pregnant, nursing mothers, or planning to become pregnant during the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-02-06 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of hMAP3 | Day 29
  Peak plasma concentrations of hMAP3 after topical application of SB414

SECONDARY OUTCOMES:
Safety Profile (Reported Adverse Events) | Day 29
  Reported Adverse Events
Subject Assessment of Tolerability | Baseline, Week 2 and Week 4
  Subject-reported from 5-point tolerability scale overall presence and degree of itching and burning/stinging
Efficacy Assessed by Target Plaque Severity Score (TPSS) | Baseline, Week 2 and Week 4
  Target Plaque Severity Score will be collected
Pharmacodynamics of SB414 | Day 29
  Change in relevant Pre and Post-dose tissue cytokine levels (mg/mg tissue)
Efficacy Assessed by Physician's Static Global Assessment | Screening, Baseline, Week 2 and Week 4
  Physician's Static Global Assessment based on overall evaluation of the disease severity
Efficacy as assessed by Itch Numeric Rating Scale (NRS) | Screening, Baseline, Week 2 and Week 4
  Itching due to psoriasis as reported by subject on a 11-point rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Tomoko Maeda-Chubachi, MD, Study Chair — Novan, Inc.
Locations (4):
- United States (4):
  - Novella Site# 247, Boise, Idaho
  - Novella Site# 183, Austin, Texas
  - Novella Site# 249, College Station, Texas
  - Novella Site# 114, Norfolk, Virginia